CLINICAL TRIAL: NCT01354977
Title: Effect of Resveratrol on Age-related Insulin Resistance and Inflammation in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Meredith Hawkins, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-534
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Diabetes Mellitus; Endocrine System Diseases; Resveratrol; Therapeutic Uses
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Diseases; Diabetes Mellitus; Endocrine System Diseases | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Resveratrol (Experimental): Each participant will receive a 28 days' supply of resveratrol capsules on day 0.
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — 1,000mg twice daily for 28 days
  Other Names: 3,5,4'-trihydroxy-trans-stilbene

SUMMARY:
Resveratrol is a natural polyphenol (a compound containing a phenol functional group) that can be found in many plants. The purpose of this research is to study the effects of resveratrol on the action of insulin (a hormone produced in the body by the pancreas that regulates the amount of sugar in the blood), fat accumulation, and inflammation in the body.

DETAILED DESCRIPTION:
Participants will meet with the study team to discuss dietary recommendations. Each participant will be instructed to follow a standardized diet plan and to avoid vigorous exercise before beginning the study. Participants will be given a 28 day supply of resveratrol capsules (Two 500 mg capsules taken twice a day). A comprehensive study of whole-body insulin action called a pancreatic clamp will be done and small samples of fat and muscle will be taken before and after the administration of resveratrol.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 26-35
* Non-smoker
* Normal screening labs (CMC, chemistry, LFTs PT/PTT)
* No CAD
* Good IV access

Exclusion Criteria:

* High cholesterol
* <4 week history of participation in another drug trial
* Severe hypertension
* Heart disease
* Liver disease of liver abnormalities
* Cerebrovascular disease, i.e. stroke
* CVD
* Seizures
* Bleeding disorders
* Muscle disease
* Cancer
* HIV
* Hepatitis (all types)
* Mentally disabled persons
* Pregnant women
* Allergies to Novocaine, Lidocaine, Benzocaine
* Subjects on the following medications:

  * Anticoagulant and antiplatelet drugs
  * Anti-epileptic drugs
  * Mexiletene
  * Quinidine
  * Cyclosporine
  * Tacrolimus
  * HIV protease inhibitors

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith A Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Resveratrol: Each participant received resveratrol, 1,000mg twice daily for 28 days in a randomized, double blinded placebo-controlled fashion.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of Resveratrol. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
- Placebo: Each participant received a supply of placebo (similar in taste and appearance to Resveratrol) twice daily for 28 days in a randomized, double blinded placebo-controlled fashion.
  The investigators used a research procedure called a "pancreatic clamp" study to study the effects of Resveratrol. During the clamp procedure, glucose (a sugar) and insulin (a hormone that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism.
Period: Overall Study
Arm/Group | Resveratrol | Placebo
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We administered a dose of 2 gm/day Resveratrol (RV) or placebo (PL) for 28 days in a randomized, double-blinded study to total of 20 non-diabetic subjects.
Groups:
- Resveratrol: Each participant received a supply of resveratrol (1,000mg) twice daily for 28 days
- Placebo: Each participant received a supply of placebo (similar in taste and appearance to Resveratrol) twice daily for 28 days
- Total: Total of all reporting groups
Arm/Group | Resveratrol | Placebo | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.75 (10.50) | 52.88 (5.44) | 51.6 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 2 | 3
  Ethnicity: Not Hispanic or Latino | 11 | 6 | 17
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Insulin Sensitivity (RD) Measured by the Change in Glucose Rates of Disappearance With Resveratrol or Placebo at Baseline and at 4 Weeks.
Description: We will measure peripheral insulin sensitivity by determining the rate of glucose uptake (RD).
  RD will be measured using a 6 hours stepped pancreatic clamp study procedure under various treatment conditions (eg, resveratrol or placebo). by monitoring changes in the level of a non-radioactive, naturally occurring form of glucose (sugar).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 12 | 8
mg/kg/min
  RD at baseline | 6.573 (1.709) | 7.272 (2.810)
  RD at 4 weeks | 8.445 (3.616) | 7.419 (2.785)

2. Secondary Outcome: Endogenous Glucose Production (EGP), With Resveratrol or Placebo at Baseline and at 4 Weeks.
Description: Endogenous glucose production will be used to determine hepatic insulin sensitivity.
  Rates of EGP (a measure of the body's production of sugar) will be measured using a 6 hour stepped pancreatic clamp procedure under various treatment conditions (eg, resveratrol or placebo), by monitoring changes in the level of a non-radioactive, naturally occurring form of glucose (sugar).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 12 | 8
mg/kg/min
  EGP at baseline | 1.014 (0.353) | 0.903 (0.436)
  EGP at 4 weeks | 1.140 (0.525) | 1.552 (0.962)

3. Secondary Outcome: Effects of Resveratrol on Skeletal Muscle Mitochondrial Numbers
Description: Skeletal muscle mitochondria numbers were calculated under EM on subjects pre- and post- treatment of either Resveratrol or placebo intervention.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mitochondria number
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 12 | 8
mitochondria number
  Baseline_mitochondria number | 48.489 (13.180) | 41.275 (10.826)
  4 weeks_mitochondria number | 46.622 (18.895) | 48.850 (14.632)

4. Secondary Outcome: Gene Expression in Whole Fat Tissue , Before and After 4 Weeks' Resveratrol and Placebo. Ratio From Baseline Versus at 4 Weeks
Description: Changes of relative copy number of gene inflammatory markers in whole fat tissue were studied by quantitative, real-time RT-PCR, resveratrol vs. placebo
Time Frame: 4 weeks
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 12 | 8
Ratio
  TNFa_Whole adipose tissue | 0.47 (0.21) | 1.4 (0.82)
  IL6_Whole adipose tissue | 1.84 (3.59) | 1.68 (1.3)
  PAI-1_Whole adipose tissue | 0.56 (0.16) | 0.76 (0.25)

5. Secondary Outcome: Muscle Mitochondrial Area
Description: Skeletal Muscle Mitochondria Area Before and After 4 Weeks of Resveratrol/Placebo Treatment
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: µm²
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 12 | 8
µm²
  Baseline_mitochondria area | 0.070 (0.021) | 0.080 (0.026)
  4 weeks_mitochondria area | 0.098 (0.039) | 0.102 (0.020)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 weeks.
Description: Not reported
Arm/Group | Resveratrol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 3/12 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol (N=12) | Placebo (N=8)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphoresis, nausea and lightheadedness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vasovagal reflex (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT01354977/Prot_SAP_000.pdf